CLINICAL TRIAL: NCT00732316
Title: HLA-HAPLOIDENTICAL FAMILIAL DONOR HEMATOPOIETIC CELL TRANSPLANTATION AFTER REDUCED INTENSITY CONDITIONING OF BUSULFAN, FLUDARABINE, AND ANTI-THYMOCYTE GLOBULIN FOR ADULT PATIENTS WITH HEMATOLOGIC MALIGNANCIES AND MYELODYSPLASTIC SYNDROME - A PHASE 2 STUDY
Brief Title: Donor Stem Cell Transplant After Busulfan, Fludarabine, and Antithymocyte Globulin in Treating Patients With Hematologic Cancer or Myelodysplastic Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Collaborators: Pusan National University Hospital (Other)
Responsible Party: Principal Investigator, Kyoo-Hyung Lee, Professor of Internal Medicine, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000600347; AMC-UUCM-2008-0037
Record Dates: First submitted 2008-08-08; First posted 2008-08-11 (Estimated); Last update posted 2012-07-17 (Estimated); Status verified 2012-07

CONDITIONS: Leukemia; Myelodysplastic Syndromes
Keywords: accelerated phase chronic myelogenous leukemia; adult acute lymphoblastic leukemia in remission; adult acute myeloid leukemia in remission; acute undifferentiated leukemia; blastic phase chronic myelogenous leukemia; childhood acute lymphoblastic leukemia in remission; childhood acute myeloid leukemia in remission; childhood chronic myelogenous leukemia; childhood myelodysplastic syndromes; chronic phase chronic myelogenous leukemia; chronic myelomonocytic leukemia; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; recurrent childhood acute lymphoblastic leukemia; recurrent childhood acute myeloid leukemia; recurrent adult acute lymphoblastic leukemia; recurrent adult acute myeloid leukemia; refractory anemia with excess blasts; refractory anemia with excess blasts in transformation; relapsing chronic myelogenous leukemia; secondary myelodysplastic syndromes
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes; Leukemia, Myeloid, Accelerated Phase; Leukemia, Biphenotypic, Acute; Blast Crisis; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myelomonocytic, Chronic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Anemia, Refractory, with Excess of Blasts | interventions — Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: nonmyeloablative allogeneic hematopoietic stem cell transplantation — administration of conditioning therapy including immunosuppressive agents plus alkylating agents and infusing hematopoietic progenitor cells collected from the donor
Procedure: peripheral blood stem cell transplantation — infusion of donor hematopoietic cells collected by leukapheresis after mobilization with growth factor

SUMMARY:
RATIONALE: Giving low doses of chemotherapy and antithymocyte globulin before a donor stem cell transplant helps stop the growth of cancer and abnormal cells. It may also stop the patient's immune system from rejecting the donor's stem cells. The donated stem cells may replace the patient's immune cells and help destroy any remaining cancer and abnormal cells (graft-versus-tumor effect).

PURPOSE: This phase II trial is studying how well a donor stem cell transplant works after busulfan, fludarabine, and antithymocyte globulin in treating patients with hematologic cancer or myelodysplastic syndrome.

DETAILED DESCRIPTION:
OBJECTIVES:

* To evaluate the efficacy of HLA-haploidentical familial donor hematopoietic cell transplantation with a reduced-intensity conditioning regimen of busulfan, fludarabine phosphate, and anti-thymocyte globulin in patients with hematologic malignancies or myelodysplastic syndromes.

OUTLINE: Before receiving the reduced-intensity conditioning regimen, patients receive one dose of intrathecal (IT) methotrexate, then leucovorin calcium IV or orally 4 hours after methotrexate and every 6 hours for a total of 8 doses.

* Reduced-intensity conditioning regimen: Patients receive busulfan IV over 6 hours on days -7 and -6, fludarabine phosphate IV over 30 minutes on days -7 to -2, anti-thymocyte globulin (ATG) IV over 4 hours on days -4 to -1, and methylprednisolone IV over 30 minutes on days -4 to -1.
* HLA-haploidentical familial donor hematopoietic stem cell transplantation (HSCT): Patients undergo allogeneic HSCT over 1 hour on days 0 and 1.
* Graft-versus-host disease (GVHD) prophylaxis: Patients receive cyclosporine IV* over 2-4 hours every 12 hours on days -1 to 30 followed by a taper until day 60 and methotrexate IV on days 2, 4 , 7, and 12.

NOTE: *Cyclosporine can be given orally once oral medication can be tolerated

* CNS prophylaxis: When blood counts recover, patients with acute leukemia or chronic myelogenous leukemia in blastic crisis resume IT methotrexate once every 2 weeks for a total of 4 doses (including the dose given before the conditioning regimen) and leucovorin calcium IV or orally 4 hours after (each dose of methotrexate) and every 6 hours for a total of 8 doses.

After completion of study treatment, patients are followed periodically for up to 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of 1 of the following hematological malignancies:

  * Acute leukemia, including any of the following:

    * Refractory acute leukemia
    * Acute leukemia beyond first remission
    * Acute leukemia in first remission with intermediate to poor prognostic features as suggested by chromosomal findings
  * Chronic myelogenous leukemia (CML)

    * Second chronic phase
    * Accelerated phase
    * Blastic phase
  * Myelodysplastic syndrome (MDS)

    * High-risk MDS (refractory anemia with excess blasts [RAEB], RAEB in transformation, and chronic myelomonocytic leukemia) can be transplanted without prior therapy or after prior therapy failure with hypomethylating agents
    * Low-risk MDS can be considered for transplantation after prior therapy failure with immunosuppressive or hypomethylating agents
* No willing, suitable HLA-matched donor in family or in donor registries

  * Patients with active hematologic malignancy, who are felt to be in urgent need of allogeneic hematopoietic cell transplantation, can enroll without a search for HLA-matched unrelated donors
* Related donor with HLA-haploidentical mismatch at 3 or less of 6 loci available

PATIENT CHARACTERISTICS:

* Karnofsky performance status 70-100%
* Bilirubin < 2.0 mg/dL
* Creatinine < 2.0 mg/dL
* AST < 3 times upper limit of normal
* Ejection fraction > 40% by MUGA

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2008-04; Primary Completion 2009-12 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
tumor response | about 4-8 weeks after transplantation
  leukemia CR, CR duration

SECONDARY OUTCOMES:
Donor cell engraftment (neutrophil, platelet, and red blood cells) | 10-35 days after transplantation
  neutrophi count over 500/ul
Acute and chronic graft-versus-host disease | 15-100 days; 100 days to 4 years
  ocurrence of acute or chronic GVHD

CONTACTS AND LOCATIONS:
Overall Officials: Kyoo H. Lee, MD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center - University of Ulsan College of Medicine, Seoul, South Korea

REFERENCES:
- [Result] Lee KH, Lee JH, Lee JH, Kim DY, Seol M, Lee YS, Kang YA, Jeon M, Hwang HJ, Jung AR, Kim SH, Yun SC, Shin HJ. Reduced-intensity conditioning therapy with busulfan, fludarabine, and antithymocyte globulin for HLA-haploidentical hematopoietic cell transplantation in acute leukemia and myelodysplastic syndrome. Blood. 2011 Sep 1;118(9):2609-17. doi: 10.1182/blood-2011-02-339838. Epub 2011 Jun 28. PMID 21715313